CLINICAL TRIAL: NCT00636116
Title: A Comparison of Anavip® and CroFab® in the Treatment of Patients With Crotalinae Envenomation: A Randomized, Prospective, Blinded, Controlled, Comparative, Multicenter Study
Brief Title: Phase 3 Multicenter Comparative Study to Confirm Safety and Effectiveness of the F(ab)2 Antivenom Anavip.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Bioclon S.A. de C.V. (Industry)
Collaborators: Universidad Nacional Autonoma de Mexico (Other); University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YA-07/02; NCT00884156 (obsolete NCT alias)
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Snake Bite
Keywords: snake bite; antivenin treatment
MeSH Terms: conditions — Snake Bites | interventions — anavip; Crotalidae Polyvalent immune Fab; Red Meat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Anavip with Anavip Maintenance Therapy
  Interventions: Biological: Crotalinae (pit viper) equine immune F(ab)2
- Group 2 (Experimental): Anavip with Placebo Maintenance Therapy
  Interventions: Biological: Crotalinae (pit viper) equine immune F(ab)2
- Group 3 (Active Comparator): CroFab with CroFab Maintenance Therapy
  Interventions: Biological: Crotalidae Polyvalent Immune Fab, ovine

INTERVENTIONS:
Biological: Crotalinae (pit viper) equine immune F(ab)2 — Anavip with Anavip Maintenance Therapy
  Other Names: Anavip
  Arms: Group 1
Biological: Crotalinae (pit viper) equine immune F(ab)2 — Anavip with Placebo Maintenance Therapy
  Other Names: Anavip
  Arms: Group 2
Biological: Crotalidae Polyvalent Immune Fab, ovine — CroFab with CroFab Maintenance Therapy
  Other Names: CroFab
  Arms: Group 3

SUMMARY:
The purpose of this study is to establish if F(ab)2 antivenom (Anavip) is safe for crotalinae envenomation. Confirm its effectiveness in preventing the occurrence of delayed coagulopathies and compare the safety and efficacy with Fab antivenom (CroFab) in patients with Crotalinae envenomation.

DETAILED DESCRIPTION:
Fewer than 200,000 crotaline envenomations occur annually in the US.Crotaline venoms contain a broad variety of toxins, venom variability and injection quantity among individual snakes and across species result in broadly variable patient presentations. Clinical consequences of crotaline envenomation include local and systemic effects, both of which may progress for hours to days.The best studied systemic consequence is coagulopathy, which may in its complexity mimic disseminated intravascular coagulation. Platelet and clotting disorders respond rapidly to administration of polyvalent antivenom.

Crotaline viper envenomation in the United States is treated with one of two licensed products: Wyeth Antivenin (Crotalidae) Polyvalent (Polyvalent), or CroFab® (antivenin Crotalidae polyvalent immune Fab, ovine). In recent years, both of these products have been in critically short supply. Use of Wyeth Polyvalent has been associated with a greater than 75% incidence of adverse reactions, including acute type 1 and delayed type 2 immune reactions.These phenomena are an inherent risk in the use of whole immunoglobulin. CroFab´s low molecular weight creates a pharmacokinetic mismatch with crotaline venom which leds to a recurrent venom effects.

Anavip is pharmacologically and pharmacokinetically different.Because of the elimination of the Fc portion of the immunoglobulin molecule, Anavip is expected to produce far fewer adverse reactions than seen with whole immunoglobulin antivenoms and unlike Fab molecules, F(ab)2 molecules exceed the size threshold for renal clearance and thus are expected to remain in circulation for a significantly longer time and substantially reduce the incidence of recurrent coagulopathy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 2 to 80 years of age
* Presenting for emergency treatment of pit viper bite
* Informed consent document read and signed by patient (or parent/legal guardian)

Exclusion Criteria:

* Current use of any antivenom, or use within the last month
* Current participation in a clinical drug study, or participation within the last month
* Positive urine or blood pregnancy test at screening
* Breast-feeding
* Allergy to horse serum, sheep serum, or papaya
* Underlying medical conditions that significantly alter platelet count or fibrinogen; thrombocytopenia, hemophilia, familial dysfibrinogenemia, leukemia
* Use of any medication expected to affect platelet count, coagulation factors or fibrinogen: chemotherapeutic agents, warfarin, heparin
* No clinical indications of snake bite requiring antivenom for treatment

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2008-05; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Incidence rate of patients experiencing coagulopathy during the follow-up phase of the study. Absolute Platelet levels < 150,000/mm3. Absolute Fibrinogen levels < 150 mg/dL. Clinical coagulopathy requiring additional antivenom. | Study Day 5 (±/- 1 day), Study Day 8 (±/- 1 day)

SECONDARY OUTCOMES:
Comparison between groups of: Percentage of patients who experience venonemia. Absolute platelet level measured Lowest absolute platelet level measured Absolute fibrinogen level Lowest absolute fibrinogen level | Study Day 5 (+/- 1 day) and Study Day 8 (+/- 1 day)

CONTACTS AND LOCATIONS:
Overall Officials: Walter García Ubbelohde, MD, Study Director — Instituto Bioclon
Locations (18):
- United States (18):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Maricopa Integrated Health System, Phoenix, Arizona
  - Northwest Medical Center, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - University Physicians Hospital, Tucson, Arizona
  - University Medical Center, Tucson, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - University of California San Diego, San Diego, California
  - Rady Children's Hospital, San Diego, California
  - Florida Poison Information Center, Jacksonsville, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - LSU Health Sciences Center, Lousiana Poison Control Center, Shreveport, Louisiana
  - The Children's Mercy Hospital, Kansas City, Missouri
  - The University of New Mexico Hospital, Albuquerque, New Mexico
  - Pitt County Memorial Hospital, Greenville, North Carolina
  - St. Joseph Regional Health Center, Bryan, Texas
  - West Texas Regional Poison Center at Thomason Hospital, El Paso, Texas
  - Scott and White Memorial Hospital, Temple, Texas